# The Steno Tech Explore study – research protocol

# **Contents**

| 0. | Cover page | 2 |
|----|-------------------------------------------|---|
| | Introduction | |
| | Aim | |
| | Methods | |
| | 3.1 Study groups/cohorts | |
| | 3.2 Participant eligibility and selection | |
| | 3.3 Survey recruitment procedure | |
| | 3.4 Data collection procedure | |
| | 3.5 Survey content | |
| | 3.6 Register and EMR data | |
| | 3.7 Data analysis | |
| | 3.8 Ethics | |
| | Results | |
| | References | |
| | Appendices | |
| | 6.1 Appendix 1: The Steno Tech Survey | |
| | 11 | |

# 0. Cover page

**Official title:** Steno Tech Explore: A Multisite Exploratory Study of People with Type 1 Diabetes on Insulin Pump Therapy

NTC number: NCT04311164

Document date: January 22, 2021

#### 1. Introduction

Optimal diabetes self-management in people with type 1 diabetes is important to minimize the risk of developing long-term microvascular and macrovascular complications (1, 2). However, only 21% of US adults with type 1 diabetes achieve the recommended target glycated hemoglobin level (HbA1c) of < 7.0% (53 mmol/mol) (3) and recent Danish data show success rates of approximately 25% (4).

One way to improve self-management and thus prevent or delay complications is to introduce diabetes technologies such as continuous subcutaneous insulin infusion (CSII) and/or continuous glucose monitoring (CGM) into individuals' treatment regimens. An estimated 40-62% of adults with type 1 diabetes in the US and 5-15% of those in Europe use CSII with or without CGM (5). Recent observational data from the type 1 diabetes Exchange registry show that while not reaching HbA1c target on average, people using CSII achieve improved metabolic outcomes compared to people using multiple daily injections, and that combining CSII with CGM substantially improves outcomes (3). However, it is recognized that reaping the benefits of these technologies requires high levels of engagement from users and health care professionals (HCPs), and that outcomes vary greatly among individuals (6-8).

To ensure optimal use of CSII and/or CGM, it is recommended that people with type 1 diabetes receive structured and recurring education (6, 7, 9). Yet, there is currently no consensus on which educational practice is best for a given patient (9, 10), and the literature indicates a paucity of high quality comparative studies regarding the effectiveness of technology-specific education (11, 12). Studies involving technology-specific education have shown that people with type 1 diabetes treated with CSII often do not use advanced pump functions or benefit substantially (13-15). These observations are concerning, particularly when combined with findings that using advanced functions can lead to improved HbA1c (16-19). It is frequently found that device-specific satisfaction is a good predictor of device utilization (20-23); however, preferences for device properties have seldomly been investigated or linked to outcomes and treatment goals of the individual (24). Whereas research mostly has focused on device-specific preferences and satisfaction (20-24), only little research has been conducted into individuals' needs and preferences for technology-specific education (12). However, meeting the needs and integrating the preferences of the individual in new interventions is considered integral to ensuring patient-centered and effective care (25-27). Accordingly, taking the target group's needs and preferences into account is essential to developing effective educational strategies (11, 25).

There are other barriers to treatment success than acquiring and maintaining the necessary skills to successfully manage CSII. For example, factors such as age and baseline HbA1c at treatment initiation have been identified as important predictors of treatment success in CSII-users (28-33).

Only a modest amount of literature has examined how psychosocial factors predict success (34, 35), with one study finding that psychological determinants, especially self-efficacy and locus of control, account for 50% of observed variation in HbA1c in people with type 1 diabetes using CSII (34). Likewise, an important known psychosocial predictor of poor diabetes outcomes is diabetes distress. One study found that a high level of diabetes distress was associated with higher HbA1c and less time in range compared to moderate or low levels of diabetes distress in people with type 1 diabetes using CSII; however, the high diabetes distress group did not perform less pump-specific

self-management activities (e.g., use of bolus wizard) suggesting that other mechanisms than technology-specific behavior may drive differences in outcomes (36). Thus, alongside demographic, socioeconomic and health status factors, psychological and psychosocial predictors may play a significant yet underexplored part in the successful use of diabetes technology.

## 2. Aim

The present study is part of an overarching study being conducted in Denmark at Steno Diabetes Center Copenhagen (SDCC) and Nordsjællands Hospital Hillerød (NOH), Steno Tech, that aims to develop and ultimately, in a randomized controlled trial (RCT), test approaches that can assist people with type 1 diabetes in obtaining optimal outcomes using CSII. Through a large-scale, questionnaire-based online survey enriched with data from national registers, this sub-study contributes to this overarching aim by exploring the importance of individual differences across a wide range of factors, including demographic, socioeconomic, health status, psychosocial and preference structures, for optimal use of CSII in people with type 1 diabetes.

#### 3. Methods

## 3.1 Study groups/cohorts

The study population consists of two groups/cohorts:

- 1. Steno Tech Survey Respondents: A cohort of individuals with type 1 diabetes treated with CSII at either SDCC or NOH participating in the Steno Tech Survey.
- 2. General Type 1 Diabetes Population: A cohort consisting of the entire population of people with type 1 diabetes in Denmark not included in the Steno Tech Survey cohort (ca. 25.000 individuals).

### 3.2 Participant eligibility and selection

All adults (18+ years) with type 1 diabetes using CSII attending SDCC or NOH was invited to participate in the survey (N = 1,592); however, people who were not fluent in Danish were excluded as the survey was only available in Danish. The general type 1 diabetes group will be identified via the National Patient Registry (NPR) once data are ready for analysis (see section 3.6).

#### 3.3 Survey recruitment procedure

Beginning in quarter 3 of 2019, eligible survey participants were approached by their primary HCP in conjunction with a consultation at SDCC or NOH and invited to participate in the survey. If they agreed to participate, they received, upon survey-opening, an invitation in e-Boks<sup>1</sup> with a link to the survey and a standardized, mandatory document containing information on how their data would be stored and used. Before answering the survey, participants were prompted to provide written consent.

<sup>&</sup>lt;sup>1</sup> e-Boks is an electronic mailbox designed to provide a digital and secure communication path between Danish citizens, companies and public authorities. As of quarter 2 of 2019, 91.5% of all Danish citizens have an e-Boks.

### 3.4 Data collection procedure

The survey was designed and administered in REDCap, an online browser-based data and survey management tool. The REDCap server is encrypted, logged and administered by the Capital Region of Denmark. Thus, the tool is cleared for storing and handling person-sensitive information according to Danish law.

The survey data are to be merged with outcome and other input data from electronic medical records (EMRs) and national Danish registers and stored and analyzed on a secure server at Statistics Denmark (figure 1).

Figure 1: Overview of data sources



## 3.5 Survey content

The survey consisted of multiple elements as per the study aim (table 1 presents an overview, appendix 1 presents the survey in full). Importantly, this sub-study is preceded by a qualitative part of the Steno Tech Explore study that explored: 1) possibilities and barriers to effective daily insulin pump management, 2) specific circumstances and contexts in relation to the possibilities and barriers such as availability and appropriateness of structured education and other support, and 3) needs and preferences in overcoming barriers and optimizing possibilities for implementing and managing technology in daily life. The content of the survey is partly inspired by concepts and themes identified in that study and partly by systematic literature reviews (11, 12, 37, 38) and professional experience.

Table 1: Overview of survey content

| Survey parts | Single survey items | Survey questionnaire scales | Survey<br>page<br>nrs.* |
|---|---|---|---|
| 1) Insulin pump and sensor-specific characteristics and behavior | <ul> <li>▼ Type(s) of device(s)</li> <li>▼ Reason(s) for device start</li> <li>▼ Device functions used</li> <li>▼ Data upload practices</li> </ul> | Insulin Device Satisfaction Survey (IDSS)(22): consists of 13 items has three subscales: 1) perceived effectiveness, 2) burden, and 3) inconvenience. Glucose Monitoring System Satisfaction Survey (GMSS)(39): consists of 15 items and has four subscales: 1) openness, 2) emotional burden, 3) behavioral burden, 4) trust. New insulin pump attitude scale compiled of questions from validated scales(40, 41): included 8 items specifically about wearing an insulin pump (e.g., the degree to which it makes one feel less attractive) and everyday challenges (e.g., the degree to which it is a problem during sex). | 2-5, 10-12 |
| 2) Experience with insulin pump education | <ul> <li>Received education (group/individual)</li> <li>Desired education (group/individual)</li> <li>Insulin pump-knowledge and support needs</li> </ul> | | 6-8 |
| 3) Carbohydrate counting exercise | <ul> <li>Chocolate (6 images)</li> <li>Pasta (6 images)</li> <li>Grapes (6 images)</li> <li>Bread rolls (5 images)</li> </ul> | Respondents were asked to indicate if they ate the presented food items 1) never, 2) occasionally or 3) often. If occasionally or often, they were shown an image and asked to pick the serving size they would usually eat and to eyeball the amount of carbohydrates in that serving size. | 9 |
| 4) Health-management behavior | <ul> <li>Physical activity</li> <li>Diet</li> <li>Alchol intake</li> <li>Smoking status</li> </ul> | Items about physical activity, diet, alcohol intake, and smoking status were based on recommended guidelines from the Danish Health Authority. | 13 |

| 5) General and diabetes- | | Well-Being Index (WHO5)(42): consists of 5 items. | 14-16, 19- |
|---|---|---|---|
| specific psychosocial<br>health | | Hypoglycemia Fear Survey short-form (HFS-SF)(43): consists of 11 items and has a worry and a behavior subscale. | 20 |
| | | Type 1 Diabetes Distress Scale (T1-DDS)(44): consists of 28 items and has seven subscales: 1) powerlessness, 2) management distress, 3) hypoglycaemia distress, 4) negative social perceptions, 5) eating distress, 6) physician distress, and 7) friend/family distress. | |
| | | <b>DAWN Support for Diabetes Self-Management Profile (DSDSP)</b> (extended)(45): this version of the DSDSP consists of 6 items. | |
| | | <b>The COVID-19 Impact on Quality of Life Profile</b> (46): The COVID-19 Impact on Quality of Life Profile is a newly-designed scale, inspired by the 'DAWN Impact of Diabetes Profile (DIDP)' scale and consists of 9 items. | |
| 6) Personality factors and goal-setting | <ul> <li>▼ Self-efficacy</li> <li>▼ Time preferences</li> <li>▼ Risk aversion</li> <li>▼ Treatment goals</li> </ul> | General Self-Efficacy Scale (GSE)(47): consists of 10 items. | 17-18, 21-<br>27 |
| 7) Self-rated health status and satisfaction with life | <ul><li>♥ Health status VAS</li><li>♥ Life satisfaction VAS</li></ul> | Both VAS scales ranged from 0-10, with 10 respresenting the best thinkable health status/satisfaction and 0 the worst. | 19 |

Abbreviations: N/A = not applicable; VAS = visual analog scale. \*Page numbers refer to actual order in the survey and correspond to appendix XX including all survey items.

#### 3.6 Register and EMR data

Register data will be obtained via Statistics Denmark and include variables from several registers, including the following population registries: The National Population Registry, the Civil Registration System, the Education Registry, the Income Registry and the Address Registry, and the following health registries: the National Patient Registry, the National Prescription Registry, the Hospital Medicine Registry, and the Health Insurance Registry. A data extraction agreement with Statistics Denmark has been made and is currently being processed.

Key population variables extracted for both study groups include, but are not limited to, gender, age, education, occupation and income (socioeconomic status), as well as household composition, all encounters with the health care system in the survey period (e.g., if the participant has been admitted to the hospital with a ketoacidosis), redeemed prescriptions from hospitals and pharmacies, and distance to health care services from private address.

Diabetes-specific clinical outcomes in both study groups will be extracted from registers, and from survey respondents' EMRs. Register-extracted outcomes include all blood and urine test measures taken at the annual 'check-up', including HbA1c, hemoglobin, eGFR, UACR, cholesterol total, HDL, LDL, VLDL, triglycerides, diabetes-related complications and other somatic and psychiatric comorbidities. EMR-extracted outcomes (available only for the survey group) include BMI, blood pressure and hypoglycemia awareness status, which are not tracked in national registers.

#### 3.7 Data analysis

The overall data analysis approach is based on descriptive, non-parametric and parametric statistical methods. Descriptive statistics will include amounts/counts (n), shares (%), means and variable distributions (standard deviations and percentiles). Non-parametric hypothesis tests will include the Chi-squared test, Fisher's exact test and Wilcoxon rank test depending on variable distributions. Parametric hypothesis tests will center on Student's unpaired and paired t-tests as well as general and generalized regression analyses. Model error structures will depend on the specific objective but, in general, take the following form:

$$Y_i = \beta_0 + \beta_1 X_{1i} + \beta_2 X_{2i} + \dots + \beta_n X_{ni} + e_i$$

where Y is the dependent variable (e.g., HbA1c) for individual i,  $\beta_n$  is the effect on  $Y_i$  given  $X_n$ , where  $X_n$  indicates demographic, socioeconomic, behavioral and psychosocial factors, and  $e_i$  indicates residual error (i.e., unexplained variance).

Furthermore, quasi-experimental procedures such as propensity score or coarsened exact matching and machine-learning algorithms such as random forest will be employed to maximize data usage and to foster meaningful comparisons within and between the two study groups.

#### 3.8 Ethics

The study was approved by the Danish Data Protection Agency (P-2019-812) and exempted from review by the Capital Region of Denmark's Research Ethics Committee (19080899). The study was also registered on ClinicalTrials.gov (NCT04311164).

# 4. Results

Data collection for this study is currently in progress. Survey data collection was initiated on May 15, 2020 and completed on October 15, 2020. In total, 770 individuals responded to the survey. EMR and register data are currently being extracted and prepared for merge with survey data by Statistics Denmark.

#### 5. References

- 1. Diabetes C, Complications Trial Research G, Nathan DM, Genuth S, Lachin J, Cleary P, et al. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. *N Engl J Med* 1993; **329**: 977-986.
- 2. Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, et al. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. *N Engl J Med* 2005; **353**: 2643-2653.
- 3. Foster NC, Beck RW, Miller KM, Clements MA, Rickels MR, DiMeglio LA, et al. State of Type 1 Diabetes Management and Outcomes from the T1D Exchange in 2016-2018. *Diabetes Technol Ther* 2019; **21**: 66-72.
- 4. Dansk Voksen Diabetes Database, Dansk Register for Børne- og Ungdomsdiabetes, Landsdækkende klinisk kvalitetsdatabase for screening af diabetisk retinopati og maculopati, Regionernes Kliniske Kvalitetsudviklingsprogram. Dansk Diabetes Database National årsrapport 2017/2018. Copenhagen, Denmark 2018.
- 5. Naranjo D, Tanenbaum ML, Iturralde E, Hood KK. Diabetes Technology: Uptake, Outcomes, Barriers, and the Intersection With Distress. *J Diabetes Sci Technol* 2016; **10**: 852-858.
- 6. Franklin V. Influences on Technology Use and Efficacy in Type 1 Diabetes. *J Diabetes Sci Technol* 2016; **10**: 647-655.
- 7. Barnard KD, Breton MD. Diabetes Technological Revolution: Winners and Losers? *J Diabetes Sci Technol* 2018; **12**: 1227-1230.
- 8. Pickup JC. Is insulin pump therapy effective in Type 1 diabetes? *Diabet Med* 2019; **36**: 269-278.
- 9. Grunberger G, Abelseth JM, Bailey TS, Bode BW, Handelsman Y, Hellman R, et al. Consensus Statement by the American Association of Clinical Endocrinologists/American College of Endocrinology insulin pump management task force. *Endocr Pract* 2014; **20**: 463-489.
- 10. Pickup JC. The evidence base for diabetes technology: appropriate and inappropriate metaanalysis. *J Diabetes Sci Technol* 2013; 7: 1567-1574.
- 11. Jayasekara RS, Munn Z, Lockwood C. Effect of educational components and strategies associated with insulin pump therapy: a systematic review. *Int J Evid Based Healthc* 2011; **9**: 346-361.
- 12. Payk M, Robinson T, Davis D, Atchan M. An integrative review of the psychosocial facilitators and challenges of continuous subcutaneous insulin infusion therapy in type 1 diabetes. *J Adv Nurs* 2018; **74**: 528-538.
- 13. Group RS. Relative effectiveness of insulin pump treatment over multiple daily injections and structured education during flexible intensive insulin treatment for type 1 diabetes: cluster randomised trial (REPOSE). *BMJ* 2017; **356**: j1285.
- 14. Ehrmann D, Kulzer B, Schipfer M, Lippmann-Grob B, Haak T, Hermanns N. Efficacy of an Education Program for People With Diabetes and Insulin Pump Treatment (INPUT): Results From a Randomized Controlled Trial. *Diabetes Care* 2018; 41: 2453-2462.
- 15. Joubert M, Morera J, Vicente A, Rod A, Parienti JJ, Reznik Y. Cross-sectional survey and retrospective analysis of a large cohort of adults with type 1 diabetes with long-term continuous subcutaneous insulin infusion treatment. *J Diabetes Sci Technol* 2014; **8**: 1005-1010.
- 16. Mameli C, Scaramuzza AE, Ho J, Cardona-Hernandez R, Suarez-Ortega L, Zuccotti GV. A 7-year follow-up retrospective, international, multicenter study of insulin pump therapy in children and adolescents with type 1 diabetes. *Acta Diabetol* 2014; **51**: 205-210.
- 17. Cukierman-Yaffe T, Konvalina N, Cohen O. Key elements for successful intensive insulin pump therapy in individuals with type 1 diabetes. *Diabetes Res Clin Pract* 2011; **92**: 69-73.
- 18. Walsh J, Roberts R, Bailey T. Guidelines for optimal bolus calculator settings in adults. *J Diabetes Sci Technol* 2011; **5**: 129-135.

- 19. O'Connell MA, Donath S, Cameron FJ. Poor adherence to integral daily tasks limits the efficacy of CSII in youth. *Pediatr Diabetes* 2011; **12**: 556-559.
- 20. Walsh J, Roberts R, Weber D, Faber-Heinemann G, Heinemann L. Insulin Pump and CGM Usage in the United States and Germany: Results of a Real-World Survey With 985 Subjects. *J Diabetes Sci Technol* 2015; **9**: 1103-1110.
- 21. Peyrot M, Rubin RR. Patient-reported outcomes for an integrated real-time continuous glucose monitoring/insulin pump system. *Diabetes Technol Ther* 2009; **11**: 57-62.
- 22. Polonsky WH, Fisher L, Hessler D, Edelman SV. Development of a New Measure for Assessing Insulin Delivery Device Satisfaction in Patients with Type 1 and Type 2 Diabetes. *Diabetes Technol Ther* 2015; **17**: 773-779.
- 23. Heinemann L, Freckmann G, Ehrmann D, Faber-Heinemann G, Guerra S, Waldenmaier D, et al. Real-time continuous glucose monitoring in adults with type 1 diabetes and impaired hypoglycaemia awareness or severe hypoglycaemia treated with multiple daily insulin injections (HypoDE): a multicentre, randomised controlled trial. *Lancet* 2018; **391**: 1367-1377.
- 24. Perard R, Orme M. A Discrete Choice Experiment to Evaluate Blood Glucose Meter Preferences in People with Type 1 and Type 2 Diabetes in the UK. *Intern Med* 2014; **S6**: S6:008.
- 25. Fan L, Sidani S. Preferences of Persons with Type 2 Diabetes for Diabetes Self-Management Education Interventions: An Exploration. *Health* 2017; **9**: 1569-1588.
- 26. Sidani S, Epstein D, Miranda J. Eliciting patient treatment preferences: A strategy to integrate evidence-based and patient-centered care. *Worldviews Evid Based Nurs* 2006; **3**: 116-123.
- 27. Sidani S, Miranda J, Epstein D, Fox M. Influence of treatment preferences on validity: a review. *Can J Nurs Res* 2009; **41**: 52-67.
- 28. Shalitin S, Gil M, Nimri R, de Vries L, Gavan MY, Phillip M. Predictors of glycaemic control in patients with Type 1 diabetes commencing continuous subcutaneous insulin infusion therapy. *Diabet Med* 2010; **27**: 339-347.
- 29. Clements M, Matuleviciene V, Attvall S, Ekelund M, Pivodic A, Dahlqvist S, et al. Predicting the effectiveness of insulin pump therapy on glycemic control in clinical practice: a retrospective study of patients with type 1 diabetes from 10 outpatient diabetes clinics in Sweden over 5 years. *Diabetes Technol Ther* 2015; **17**: 21-28.
- 30. Jankovec Z, Cesak V, Krcma M, Zourek M, Rusavy Z. Can we predict success of insulin pump therapy? *J Diabetes* 2014; **6**: 384-386.
- 31. Neylon OM, O'Connell MA, Skinner TC, Cameron FJ. Demographic and personal factors associated with metabolic control and self-care in youth with type 1 diabetes: a systematic review. *Diabetes Metab Res Rev* 2013; **29**: 257-272.
- 32. Neylon OM, Skinner TC, O'Connell MA, Cameron FJ. A novel tool to predict youth who will show recommended usage of diabetes technologies. *Pediatr Diabetes* 2016; **17**: 174-183.
- 33. Andersen HU, Hangaard S, Hommel E, Ridderstrale M. Six-Year Follow-Up After Insulin Pump Initiation: HbA1c Is Significantly Reduced Without Weight Gain. *J Diabetes Sci Technol* 2018; **12**: 535-536.
- 34. Aberle I, Scholz U, Bach-Kliegel B, Fischer C, Gorny M, Langer K, et al. Psychological aspects in continuous subcutaneous insulin infusion: a retrospective study. *J Psychol* 2009; **143**: 147-160.
- 35. Indelicato L, Mariano V, Galasso S, Boscari F, Cipponeri E, Negri C, et al. Influence of health locus of control and fear of hypoglycaemia on glycaemic control and treatment satisfaction in people with Type 1 diabetes on insulin pump therapy. *Diabet Med* 2017; **34**: 691-697.
- 36. Khan A, Choudhary P. Investigating the Association Between Diabetes Distress and Self-Management Behaviors. *J Diabetes Sci Technol* 2018; **12**: 1116-1124.

- 37. Madsen KP, Kjaer T, Skinner T, Willaing I. Time preferences, diabetes self-management behaviours and outcomes: a systematic review. *Diabet Med* 2019; **36**: 1336-1348.
- 38. Grose DN, O'Brien CL, Castle DJ. Type 1 diabetes and an insulin pump: an iterative review of qualitative literature. *Practical Diabetes* 2017; **34**: 281-287.
- 39. Polonsky WH, Fisher L, Hessler D, Edelman SV. Development of a New Measure for Assessing Glucose Monitoring Device-Related Treatment Satisfaction and Quality of Life. *Diabetes Technol Ther* 2015; **17**: 657-663.
- 40. Bergis D, Roos T, Ehrmann D, Schmitt A, Schipfer M, Haak T, et al. Perceived Benefits and Barriers Regarding CSII Treatment: Development and Psychometric Evaluation of the Insulin Pump Attitudes Questionnaire (IPA-Questionnaire). *Exp Clin Endocrinol Diabetes* 2019.
- 41. Tanenbaum ML, Hanes SJ, Miller KM, Naranjo D, Bensen R, Hood KK. Diabetes Device Use in Adults With Type 1 Diabetes: Barriers to Uptake and Potential Intervention Targets. *Diabetes Care* 2017; **40**: 181-187.
- 42. Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. *Psychother Psychosom* 2015; **84**: 167-176.
- 43. Grabman J, Vajda Bailey K, Schmidt K, Cariou B, Vaur L, Madani S, et al. An empirically derived short form of the Hypoglycaemia Fear Survey II. *Diabet Med* 2017; **34**: 500-504.
- 44. Fisher L, Polonsky WH, Hessler DM, Masharani U, Blumer I, Peters AL, et al. Understanding the sources of diabetes distress in adults with type 1 diabetes. *J Diabetes Complications* 2015; **29**: 572-577.
- 45. Nicolucci A, Kovacs Burns K, Holt RI, Comaschi M, Hermanns N, Ishii H, et al. Diabetes Attitudes, Wishes and Needs second study (DAWN2): cross-national benchmarking of diabetes-related psychosocial outcomes for people with diabetes. *Diabet Med* 2013; **30**: 767-777.
- 46. Holmes-Truscott E, Skovlund SE, Hendrieckx C, Pouwer F, Peyrot M, Speight J. Assessing the perceived impact of diabetes on quality of life: Psychometric validation of the DAWN2 Impact of Diabetes Profile in the second Diabetes MILES Australia (MILES-2) survey. *Diabetes Res Clin Pract* 2019; **150**: 253-263.
- 47. Mikkelsen EG, Schwarzer R, Jerusalem M. Danish Version of the General Self-Efficacy Scale. 1999.
- 48. Acquadro C, Conway K, Hareendran A, Aaronson N, European Regulatory I, Quality of Life Assessment G. Literature review of methods to translate health-related quality of life questionnaires for use in multinational clinical trials. *Value Health* 2008; **11**: 509-521.

# 6. Appendices

## 6.1 Appendix 1: The Steno Tech Survey

In the following questionnaire (see next page), the IDSS and GMSS were translated from English to Danish using the internationally recognized forward-backward translation procedure (48). Two experienced native Danish diabetes researchers fluent in English independently forward translated each scale (i.e., from English to Danish). The forward translations were then compared by a third researcher and analyzed for discrepancies, which were then discussed among all three researchers until consensus was reached. This was followed by a similar procedure, only backwards, by two other researchers, one of whom is a native English speaker fluent in Danish.

Face validity of the translated questionnaires was ensured through one-to-one interviews in the survey testing phase where, for example, the item on cost was removed from the IDSS due to irrelevance in the Danish publicly funded health care setting.

## **Steno Tech Explore survey**

Response categories

# 

Introductory page including information described in section 3.3.

Question

# 

Scale/item [branching

| logic] | | |
|---|---|---|
| The first part of the que | stionnaire is about your insulin pump usage. There | are also questions about your use |
| of sensor, if applicable. | | |
| • | vering all the questions on a page, press "next page | " at the bottom of the page in order |
| to continue. | | |
| T 1 20 . 10 . 1 | | |
| | utes to complete the entire questionnaire. You can | <u> </u> |
| - | ire later by simply shutting down the page and usin | g the link in e-Boks again – |
| disregard the "save and | What insulin pump are you currently using? | 1. MiniMed 640G |
| pumptype | You will be shown a picture of the insulin | 2. MiniMed 670G |
| | pump below when you click on the name of the | 3. MiniMed Paradigm/VEO |
| | insulin pump. | 4. Accu-Chek Combo |
| | insum pump. | 5. Accu-Chek Insight |
| | | 6. Omnipod |
| | | 7. Medtrum |
| | | 8. Tandem t:slim X2 |
| | | 9. YpsoPump |
| | | 10. Animas Vibe |
| | | 11. Other |
| | | 12. I use a hybrid closed-loop |
| | | system that I built myself with an |
| | | open-source software such as |
| | | OPENAPS, AndroidAPS or Loop. |
| pumptype_other [if | What other insulin pump are you currently | Open-ended response |
| pumptype = 11] | using? | |
| diabetesdebut | In which year were you diagnosed with type 1 | Open-ended response |
| and trouver | diabetes? If you do not remember the exact | open ended response |
| | year, please provide an approximate estimate. | |
| pumpyear | In which year did you get your first insulin | Open-ended response |
| 1 13 | pump? If you do not remember the exact year, | |
| | please provide an approximate estimate. | |
| | 1 | 1 |

| pumpindication | What was the reason that you were initially offered an insulin pump by your healthcare provider? Feel free to choose several reasons. | I had too high long-term blood glucose (HbA1c) I had major fluctuations in my blood sugar I could not feel low blood-sugars Other Do not know/do not remember |
|---|---|---|
| pumpindication_other [if pumpindication = 4] | What other reasons were behind you being offered an insulin pump? | Open-ended response |
| pumpwhy | What was(were) the reason(s) you initially agreed to use the insulin pump? Feel free to choose several reasons. | 1. To improve long-term blood glucose (HbA1c) 2. To achieve a more stable blood sugar (fewer fluctuations) 3. To reduce the number of high blood sugars 4. To reduce the number of low blood sugars 5. To get better sleep 6. To be able to eat more flexibly 7. To be able to exercise more spontaneously 8. To make it easier to take and dose insulin 9. To avoid injecting myself several times a day 10. My healthcare provider recommended it to me 11.Other insulin pump users recommended it to me 12. To make my diabetes fill less in my life 13. Other 14. Do not know/do not remember |
| pumpwhy_other [if | What other reasons were there, for you to agree | Open-ended response |
| pumpwhy = 13] | to start insulin pump treatment? | |


| Scale/item [branching logic] | Question | Response categories |
|---|---|---|
| | now you are using your current insulin p | |
| bolus | How do you usually take bolus insulin? | <ol> <li>Bolus calculator/bolus guide</li> <li>Manual bolus (including fast bolus)</li> <li>I use both equally</li> <li>I very rarely take bolus insulin</li> </ol> |
| bolus_whynot [if bolus = 4] | Why do you not typically use the bolus guide to calculate bolus insulin? | 1. It is too difficult to use 2. I did not learn it at pump start and have not started doing it since 3. I do not trust the bolus guide's calculations 4. I calculate bolus myself, as my experience is that this works best 5. Other 6. Do not know |
| bolus_whynot_other [if bolus_whynot = 5] | What other reasons are there for why you do not typically use the bolus guide to calculate bolus insulin? | Open-ended response |
| bolususe_intro [if pumptype $\neq$ 11 or 12 and bolus $\neq$ 4] | How often do you use your bolus calculator to | |
| bolususe1 [if pumptype $\neq$ 11 or 12 and bolus $\neq$ 4] | calculate bolus for food? | <ol> <li>Never/rarely</li> <li>Occasionally</li> <li>Often</li> <li>Always/almost always</li> </ol> |
| bolususe2 [if pumptype $\neq$ 11 or 12 and bolus $\neq$ 4] | calculate correction-insulin for elevated blood sugar? | <ol> <li>Never/rarely</li> <li>Occasionally</li> <li>Often</li> <li>Always/almost always</li> </ol> |
| bolusbasalfunctions_intro [if pumptype ≠ 2, 11 or 12] | How often do you use these insulin pump functions when they are relevant? [stand-alone pump users] | |
| bolus1 [if pumptype $\neq$ 2, 11 or 12 and bolus $\neq$ 4] | Combined bolus when it is relevant (e.g., for fast food) | <ol> <li>Never/rarely</li> <li>Occasionally</li> <li>Often</li> <li>Always/almost always</li> </ol> |
| bolus2 [if pumptype $\neq$ 2, 11 or 12 and bolus $\neq$ 4] | Extended bolus when it is relevant (e.g., low blood sugar before a meal) | <ol> <li>Never/rarely</li> <li>Occasionally</li> <li>Often</li> <li>Always/almost always</li> </ol> |
| basal1 [if pumptype $\neq$ 2, 11 or 12] | Temporary basal up when it is relevant (e.g., in the case of illness) | <ol> <li>Never/rarely</li> <li>Occasionally</li> <li>Often</li> <li>Always/almost always</li> </ol> |
| basal2 [if pumptype ≠ 2, 11 or 12] | Temporary basal down when it is relevant (e.g., exercise) | 1. Never/rarely 2. Occasionally 3. Often |

| | | 4. Always/almost always |
|---|---|---|
| [manuelfunctions_intro] | How often do you use these insulin | 1. I am almost never in manual |
| | pump functions when they are | mode besides when I change |
| | relevant, and you are in manual mode? | infusion set. |
| | [Medtronic 670G users] | |
| bolus1_670G [if pumptype = 2 and | Combined bolus when it is | 1. Never/rarely |
| manuelfunctions intro $\neq 1$ ] | relevant (e.g., fast food) | 2. Occasionally |
| | | 3. Often |
| | | 4. Always/almost always |
| bolus2_670G [if pumptype = 2 and | Extended bolus when it is | 1. Never/rarely |
| manuelfunctions_intro $\neq 1$ ] | relevant (e.g., low blood sugar | 2. Occasionally |
| | before a meal) | 3. Often |
| | , | 4. Always/almost always |
| basal1_670G [if pumptype = 2 and | Temporary basal up when it is | 1. Never/rarely |
| manuelfunctions_intro \neq 1] | relevant (e.g., in the case of illness) | 2. Occasionally |
| _ , , | , | 3. Often |
| | | 4. Always/almost always |
| basal2_670G [if pumptype = 2 and | Temporary basal down when it is | 1. Never/rarely |
| manuelfunctions_intro \neq 1] | relevant (e.g., exercise) | 2. Occasionally |
| _ , , | (1.2.4) | 3. Often |
| | | 4. Always/almost always |
| autofunctions_intro [if pumptype = | How often do you use temporary | 1. Never/rarely |
| 2] | target-blood sugar when relevant (e.g., | 2. Occasionally |
| | exercise) and you are in auto-mode? | 3. Often |
| | | 4. Always/almost always |
| insulindosehow [if pumptype $\neq 2$ , | When do you typically take bolus | 1. Before the meal (10 minutes or |
| 11 or 12 and bolus $\neq$ 4] | insulin for meals? | more) |
| , , | | 2. Just before the meal |
| | | 3. During the meal |
| | | 4. After the meal |
| missedbolus [if pumptype $\neq$ 2, 11 | How often do you forget bolus insulin | 1. Never |
| or 12 and bolus $\neq 4$ ] | for meals? | 2. Once a month or less |
| , , | | 3. Once a week or less |
| | | 4. Twice a week |
| | | 5. 3-4 times a week |
| | | 6. 5-6 times a week |
| | | 7. At least once a day |
| carbhow [if pumptype $\neq$ 2, 11 or 12 | How do you typically enter | 1. I typically enter the |
| and bolus $\neq 4$ | carbohydrates into the insulin pump? | estimated/calculated amount of |
| | r r | carbohydrates |
| | | 2. I typically enter the same amount |
| | | of carbohydrates regardless of small |
| | | variations in the meal |
| | | 3. I never enter carbohydrates in the |
| | | insulin pump |
| carbhow_intro [if pumptype $\neq 2$ , 11 | How often do you do the following | 1 1 |
| or 12 and bolus $\neq$ 4 and carbhow $\neq$ | when entering carbohydrates into the | |
| 3] | insulin pump? | |
| | This does not include intake of | |
| | carbohydrates at low blood sugar or as | |
| | 1 , | <u>l</u> |

| | a preventative measure before exercise. | |
|---|---|---|
| maincourse [if pumptype $\neq$ 2, 11 or | I enter at main meals | 1. Never/rarely |
| 12 and bolus $\neq$ 4 and carbhow $\neq$ 3] | | 2. Occasionally |
| , , | | 3. Often |
| | | 4. Always/almost always |
| snack1 [if pumptype $\neq$ 2, 11 or 12 | I enter anything over 10 g | 1. Never/rarely |
| and bolus $\neq 4$ and carbhow $\neq 3$ ] | carbohydrates | 2. Occasionally |
| | | 3. Often |
| | | 4. Always/almost always |
| snack2 [if pumptype $\neq$ 2, 11 or 12 | I enter anything over 5 g carbohydrates | 1. Never/rarely |
| and bolus $\neq 4$ and carbhow $\neq 3$ ] | | 2. Occasionally |
| | | 3. Often |
| | | 4. Always/almost always |
| allmeals1 [if pumptype $\neq$ 2, 11 or | I deliberately enter more carbohydrates | 1. Never/rarely |
| 12 and bolus $\neq$ 4 and carbhow $\neq$ 3] | than the calculated amount | 2. Occasionally |
| | | 3. Often |
| | | 4. Always/almost always |
| allmeals2 [if pumptype ≠ 2, 11 or | I deliberately enter less carbohydrates | 1. Never/rarely |
| 12 and bolus $\neq$ 4 and carbhow $\neq$ 3] | than the calculated amount | 2. Occasionally |
| | | 3. Often |
| | | 4. Always/almost always |


| Scale/item [branching logic] | Question | Response categories |
|---|---|---|
| The following questions are al | bout how you use data upload from your in | isulin pump to your computer and |
| how you adjust the functions of | of your insulin pump. | |
| pumpdata | How often do you transfer data from your | 1. Never |
| | insulin pump to your computer? | 2. Once a year or less |
| | | 3. 2-5 times a year |
| | | 4. Every two months |
| | | 5. Once a month |
| | | 6. Once a week or more often |
| | | 7. Every day |
| pumpdata_why [if pumpdata | Why do you transfer data from your | 1. So that my <u>healthcare provider</u> can |
| = 3, 4, 5, 6 or 7] | insulin pump to your computer? Feel free | analyze the development of my blood |
| _ | to choose several reasons. | sugar and whether the insulin pump is |
| | | set correctly |
| | | 2. So that <u>I</u> can analyze the |
| | | development of my blood sugar and |
| | | whether the insulin pump is set |
| | | correctly |
| | | 3. Other |
| | | 4. Do not know |
| Pumpdata_why_other [if | For what other reasons do you transfer | Open-ended response |
| pumpdata_why = 3] | data from your insulin pump to your | |
| | computer? | |
| pumpdata_why [if pumpdata | Why do you never/rarely transfer data | 1. I do not own a computer |
| = 1 or 2] | from your insulin pump to your computer | 2. I did not know it was a possibility |
| | at home? Feel free to choose several | 3. I do not know how to do it |
| | reasons. | 4. Data is too hard to understand |
| | | 5. It takes too long |
| | | 6. The insulin pump program is not |
| | | compatible with my computer |
| | | 7. I prefer to keep a diabetes diary |
| | | 8. I do not find the data useful |
| | | 9. I do not like seeing my data |
| | | 10. I do not want to share my data with |
| | | an insulin pump company |
| | | 11. I do not feel the need to transfer |
| | | data at home |
| | | 12. Other |
| | | 13. Do not know |
| pumpdata_whynot_other [if | For what other reasons do you not | Open-ended response |
| pumpdata_why = 12] | transfer data from your insulin pump to | |
| | your computer? | |
| pumpadjust | Who primarily decides changes in your | 1. My healthcare provider |
| | insulin pump's basic settings? E.g., | 2. Myself |
| | carbohydrates, insulin sensitivity, basal | 3. My next of kin |
| | rates. | |

| adjustself1 [if pumpadjust = | Even though it is primarily your | 1. Yes |
|---|---|---|
| 1] | healthcare provider who decides the | 2. No |
| | settings, do you do it yourself sometimes? | |
| adjustself2 [if pumpadjust = 2 | When you adjust the basic settings of the | 1. Carbohydrate ratio |
| or adjutself1 = 1] | insulin pump yourself, which ones do you | 2. Insulin sensitivity |
| | typically adjust? Feel free to choose | 3. Basal rate |
| | several options. | 4. Insulin's duration/time of action |
| | | 5. Target blood sugar |
| daysset | How many days typically pass between | Drop-down menu from 1 to 10 days. |
| | you changing insulin needle/insulin | |
| | catheter or pod/patch? | |


| Scale/item [branching logic] [branching logic] | Question | Response categories |
|---|---|---|
| The following questions are abou | The following questions are about your possible use of sensor or flash glucose measuring device. | |
| sensor | Are you currently using a sensor or flash glucose meter? | 1. Yes<br>2. No |
| sensortype [if sensor = 1] | What sensor system do you use? You will be shown a picture of the sensor system below when you click on the name of the system. | 1. Flash Libre 2. Guardian to 640/670G insulin pump 3. Minilink to Paradigm/VEO insulin pump 4. Guardian connect 5. Dexcom (G4, G5 or G6) 6. Eversense 7. Medtrum 8. Other |
| bgmeasure_flash [if sensor = 1<br>and sensortype = 1] | How often do you typically scan your Flash Libre? (press 'menu', 'browse history' and press the down arrow to 'sensor use' on your Flash Libre to see your daily number of scans). | 1. Rarer than once a day 2. 1-3 times daily 3. 4-6 times daily 4. 7-9 times daily 5. 10 or more times a day |
| flash_who [if sensortype = 1] | Who pays for your Flash Libre? | <ol> <li>Municipality</li> <li>The hospital/region</li> <li>Out-of-pocket payment</li> <li>Do not know</li> </ol> |
| sensortype_other [if sensortype = 8] | What other sensor are you using? | Open-ended response |
| sensorstop [if sensor = 0] | Have you previously used a sensor but stopped? | 1. Yes<br>2. No |
| sensorstop_why [if sensorstop = 1] | Why did you stop using a sensor? Feel free to choose several reasons. | 1. Skin problems 2. Too many alarms 3. Technical problems (e.g., signal failure) 4. Not accurate enough 5. Annoying to wear 6. Attachment problems 7. Information overload 8. It was too difficult to understand and use the sensor values 9. Other 10. Do not know/do not remember |
| sensorstop_why_other [if sensorstop_why = 9] | What other reasons were there for you choosing to stop using a sensor? | Open-ended response |

| bgmeasure [if sensor = 0] | How often do you measure your blood | 1. Less than once a day |
|---|---|---|
| | sugar? | 2. 1-3 times daily |
| | Sugui: | 3. 4-6 times daily |
| | | 4. 7-9 times daily |
| | | 5. 10 or more times a |
| F:C 13 | 1 1:1 1:1 ( " ( ) | day |
| sensoryear [if sensor = 1] | In which year did you get your first sensor? | Open-ended reponse |
| | If you do not remember the exact year, | |
| | please provide an approximate estimate | |
| sensorindication [if sensor = 1] | What was the reason for you originally | 1. I had too high long- |
| | being offered a sensor? Feel free to choose | term blood sugar |
| | several reasons. | (HbA1c) |
| | | 2. I had severe |
| | | fluctuations in my blood |
| | | sugar levels |
| | | 3. I could not feel when I |
| | | had low blood sugar |
| | | 4. I could not make |
| | | blood sugar reading |
| | | work at work (e.g., due |
| | | to hygiene requirements) |
| | | 5. I had problems with |
| | | my fingers/hands |
| | | 6. Other |
| | | 7. Do not know/do not |
| | | remember |
| | | 8. I was not offered a |
| | | sensor. I bought it and |
| | | continue to pay for it |
| | | myself |
| . 1 | William and Control | 0 1.1 |
| sensorindication_other [if | What other reasons were there for originally | Open-ended response |
| sensorindication = 6] | being offered a sensor? | |
| whysensor [if sensor = 1] | What was the reason(s) you initially agreed | 1. To improve my long- |
| | to use the sensor? Feel free to choose | term blood sugar |
| | several reasons. | (HbA1c) |
| | | 2. To achieve a more |
| | | stable blood sugar level |
| | | (fewer fluctuations) |
| | | 3. Because I could not |
| | | feel my low blood sugar |
| | | 4. To feel more |
| | | comfortable in general |
| | | 5. I could not make |
| | | blood sugar reading |
| | | work at work (e.g., due |
| | | to hygiene requirements) |
| | | 6. I had problems with |
| | | _ |
| | | my fingers/hands |

| sensordataupload whynot [if | Why do you never/rarely transfer data from | 1. I do not have a |
|---|---|---|
| sensordataupload = 1 or 2] | your sensor to your computer at home? Feel | computer |
| | free to choose several reasons. | 2. I did not know it was a |
| | | possibility |
| | | 3. I do not know how to |
| | | do it |
| | | 4. The data are too hard |
| | | to understand |
| | | 5. It takes too long |
| | | 6. The sensor program is |
| | | not compatible with my |
| | | computer |
| | | 7. I prefer to keep a |
| | | diabetes diary |
| | | 8. I do not find the data |
| | | useful |
| | | 9. I do not like seeing |
| | | my data |
| | | 10. I do not want to |
| | | share my data with a |
| | | sensor company |
| | | 11. I do not feel the need |
| | | to transfer data at home |
| | | 12. Other |
| | | 13. Do not know |
| sensordataupload_whynot_other | What other reasons are there for you not | Open-ended response |
| [if sensordataupload_whynot = | transferring data from your sensor to your | |
| 12] | computer at home? | |
| sensorshare [if sensor = $1, 3, 4, 5,$ | Do you share sensor data with your next of | 1. Yes |
| 6 or pumptype = 12. | kin using the sensor's share function? | 2. No |
| sensorshare_who [if sensorshare | Which next of kin do you share your sensor | 1. Spouse/significant |
| = 1] | data with? Feel free to choose several | other |
| | options. | 2. Children |
| | | 3. Parents |
| | | 4. Friends |
| | | 5. Others |


| Scale/item [branching logic] | Question | Response categories |
|---|---|---|
| Think back to the teaching and | d guidance you received when you start | ed your insulin pump treatment. By this |
| | or more in which you received information | ation and guidance on insulin pump |
| treatment and the use of the in | 1 1 | |
| educationtime | Approximately how long t did the | 1. 1 day or less |
| | start-up/education last? | 2. 2-3 days |
| | | 3. 3-4 days |
| | | 4. Other |
| | | 5. Do not remember |
| education_other [if | Did the start-up/education take place | Open-ended response |
| educationtime = 4] | over a longer or shorter period? | |
| | Please be specific. | |
| educationprep | How did you prepare for the insulin | 1. I found information on the internet |
| | pump start-up? Feel free to choose | about insulin pump treatment |
| | several options. | |
| | | 2. I talked to other insulin pump users in |
| | | my network |
| | | 3. I sought out groups on social media |
| | | with insulin pump users |
| | | 4. I did not seek out special information |
| | | other than the information given to me |
| | | by my health care provider |
| | | by my nearth care provider |
| | | 5. I do not remember |
| | | 3. I do not remember |
| educationhcp | Who taught you about insulin pump | 1. Representative from a pump company |
| 1 | start-up? Feel free to choose several | 2. Dietitian |
| | options. | 3. Diabetes doctor |
| | | 4. Diabetes nurse |
| | | 5. I do not remember |
| educationt | How did the teaching take place? | 1. I received mostly group-based lessons |
| | | 2. I received mostly individual |
| | | instruction |
| | | 3. I do not remember |
| educationfam | Were your relatives invited to all or | 1. Yes |
| | part of the education? | 2. No |
| | | 3. I do not remember |
| educationgroup_intro [if | To what degree do you agree with the | |
| education = 1] | following statements? | |
| educationgroup1 [if educationt | Group education suited me well | 1. Strongly disagree |
| = 1] | | 2. Disagree |
| | | 3. Neither agree nor disagree |
| | | 4. Agree |
| | | 5. Strongly agree |

| educationgroup2 [if educationt | I appreciated talking to the other | 1. Strongly disagree |
|---|---|---|
| = 1] | participants in the group and hearing | 2. Disagree |
| 1, | about their experiences | 3. Neither agree nor disagree |
| | about their experiences | 4. Agree |
| | | 5. Strongly agree |
| educationgroup3 [if educationt | I would have preferred individual | 1. Strongly disagree |
| = 1] | education | 2. Disagree |
| - 1 ] | education | 3. Neither agree nor disagree |
| | | 4. Agree |
| | | _ |
| advection amount fife described | I found it reducible that me most of him | 5. Strongly agree |
| educationgroup4 [if educationt | I found it valuable that my next of kin | 1. Strongly disagree |
| = 1 and educationfam = 1] | could participate in all or part of the | 2. Disagree |
| | education | 3. Neither agree nor disagree |
| | | 4. Agree |
| | | 5. Strongly agree |
| educationind_intro [if education | To what degree do you agree with the | |
| = 2] | following statements? | |
| educationind1 [if education = 2] | The individual education suited me | 1. Strongly disagree |
| | well | 2. Disagree |
| | | 3. Neither agree nor disagree |
| | | 4. Agree |
| | | 5. Strongly agree |
| educationind2 [if education = 2] | I appreciated having time with | 1. Strongly disagree |
| | the teacher alone without other | 2. Disagree |
| | participants present | 3. Neither agree nor disagree |
| | | 4. Agree |
| | | 5. Strongly agree |
| educationind3 [if education = 2] | I would have preferred | 1. Strongly disagree |
| | group training with others in the | 2. Disagree |
| | same situation | 3. Neither agree nor disagree |
| | | 4. Agree |
| | | 5. Strongly agree |
| educationind4 [if education = 2 | I found it valuable that my next of kin | 1. Strongly disagree |
| and education fam = 1] | could participate in all or part of the | 2. Disagree |
| | teaching | 3. Neither agree nor disagree |
| | | 4. Agree |
| | | 5. Strongly agree |


| Scale/item [branching logic] | Question | Response categories |
|---|---|---|
| <u> </u> | re about the teaching or exchange of experience you be | ave narticinated in as an |
| The following questions are about the teaching or exchange of experience you have participated in as an experienced insulin pump user. | | |
| educationnow | Have you participated in either of these types of courses in relation to your insulin pump treatment in the past 5 years? If you have participated in both, choose the course you remember best. | Carbohydrate counting course in a group "Refresher course" experience-sharing course about insulin pump in a group |
| educationgroup2intro | To what degree do you agree with the following | 3. No, I have not participated in such courses in the last 5 years |
| educationgroupzintro | statements? | |
| educationgroup21 [educationnow = 1 or 2] | Group education suited me well | <ol> <li>Strongly disagree</li> <li>Disagree</li> <li>Neither agree nor disagree</li> <li>Agree</li> <li>Strongly agree</li> </ol> |
| educationgroup22 | I appreciated talking to the other participants in the | 1. Strongly disagree |
| [educationnow = 1 or 2] | group and hearing their experiences | <ul><li>2. Disagree</li><li>3. Neither agree nor disagree</li><li>4. Agree</li><li>5. Strongly agree</li></ul> |
| educationgroup23<br>[educationnow = 1 or 2] | I would have preferred individual education | <ol> <li>Strongly disagree</li> <li>Disagree</li> <li>Neither agree nor disagree</li> <li>Agree</li> <li>Strongly agree</li> </ol> |


| Scale/item | Question | Response categories |
|---|---|---|
| [branching | | |
| logic] | | |
| In the follow | ing we ask about your current needs for knowledge, edu | ication and experience-sharing |
| about your ir | nsulin pump. | |
| knowledge1 | Do you need a refresher or more knowledge about the | 1. No |
| | use of the different insulin pump features? | 2. Yes, to some degree |
| | | 3. Yes, very much |
| | | 4. I do not know |
| knowledge2 | Do you need sparring and experience-sharing in | 1. No |
| | relation to everyday-life with your insulin pump? | 2. Yes, to some degree |
| | Topics could be family life, sport, working life, travel, | 3. Yes, very much |
| | or the fact that you carry an insulin pump 24/7 | 4. I do not know |
| knowledge3 | Do you need more practical knowledge of the upload | 1. No |
| | and interpretation of data from your insulin pump and | 2. Yes, to some degree |
| | possible sensor? (With upload we mean transferring | 3. Yes, very much |
| | data to computer/app, e.g., blood glucose levels, sensor | 4. I do not know |
| | curves and insulin doses) | |
| knowledge4 | Do you need more knowledge and/or practical training | 1. No |
| | in how you can adjust the insulin pump settings | 2. Yes, to some degree |
| | yourself? | 3. Yes, very much |
| | | 4. I do not know |
| knowledge5 | Do you seek out knowledge about new initiatives in | 1. No |
| | insulin pump treatment on, e.g., the internet or in | 2. Yes, to some degree |
| | networks with other insulin pump users outside your | 3. Yes, very much |
| | place of treatment? | 4. I do not know |


| Scale/item [branching | Question | Response |
|---|---|---|
| logic] | | categories |
| The next questions are about carbohydrate counting. | | |
| carbcount | Do you count carbohydrates? | 1. Yes |
| | | 2. No |
| carbcount_whynot [if carbcount = 2] | Why do you not count carbohydrates? Feel free to choose several reasons. | 1. I never learned it 2. It is too much of a hassle 3. I lack training/practice in it 4. I do not feel that I need it 5. Other reasons 6. I do not know |
| carbcount_whynot_other | What other reasons are there for you not counting carbohydrates? | Open-ended |
| [if carbcount_whynot = | | response |
| 5] | | |
| carbcounthow [if | What methods do you use to count carbohydrates? Feel free to | 1. I eyeball |
| carbcount = 1] | choose several methods. | 2. I use weight |
| | | 3. I use an app |
| | | 4. I use nutrition |
| | | fact declarations |
| | | 5. I use |
| | | encyclopedias |
| | | (e.g., |
| | | carbohydrate |
| | | lists) |
| | | 6. I use Google |
| | | 7. None of the |
| 1 1 5:0 | | above |
| carbcountlearn [if | How did you learn to count carbohydrates? Feel free to choose | 1. Individual |
| carbcount = 1] | several reasons. | guidance from |
| | | dietitian |
| | | 2. Carbohydrate |
| | | counting course |
| | | 3. Self-taught |
| | | (e.g., from books, |
| | | social media or |
| | | experience- |
| | | sharing with |
| | | others) |
| | | 4. None of the |
| | | above |

| carbcount_intro | You now have the opportunity to participate in a carbohydrate counting challenge. If you eat the following food items occasionally or often, you will be shown a picture of different portion sizes for the given item. You must then pick the portion size you typically eat and state the amount of carbohydrates you think it contains. The rules are simple: you cannot use aids such as carbohydrate lists, apps, or nutrition fact declarations. The idea is that you simply respond based on your immediate assessment of carbohydrate content in each item. On the last page of the questionnaire, you can compare your response with the actual amount of carbohydrates in each food. | 1. I would like to participate 2. I do not want to take part in the challenge |
|---|---|---|
| choco1 [if carbcount = 1 | How often do you eat dark chocolate? | 1. Rarely/Never |
| and carbcount_intro = 1] | 110 w often do you cut dark enocolate: | 2. Occasionally 3. Often |
| choco2 [if choco1 = 2 or | Select the image that matches the portion size you typically eat. If | 1. Portion size A |
| 3] | you typically eat a larger or smaller portion than any of the shown, | 2. Portion size B |
| | select the image that comes closest. | 3. Portion size C |
| | | 4. Portion size D |
| | | 5. Portion size E |
| 1 25:01 1 2 | | 6. Portion size F |
| choco3 [if choco1 = 2 or 3] | A B C C F F | |
| choco4 [if choco2 ≠ .] | Type the amount of carbohydrates (in grams) that are on the image | Open-ended |
| . 1 [ ] [ ] 1 | you have selected. | response |
| pasta1 [if choco1 = 1 or | How often do you eat pasta? | 1. Rarely/Never |
| choco4 ≠ .] | | <ul><li>2. Occasionally</li><li>3. Often</li></ul> |
| pasta2 [if pasta1 = 2 or | Select the image that matches the portion size you typically eat. If | 1. Portion size A |
| 3] | you typically eat a larger or smaller portion than any of the shown, | 2. Portion size B |
| | select the image that comes closest. | 3. Portion size C |
| | | 4. Portion size D |
| | | 5. Portion size E |
| | | 6. Portion size F |

| | | , |
|---|---|---|
| pasta3 [if pasta1 = 2 or 3] | D E F | |
| pasta4 [if pasta2 ≠ .] | Type the amount of carbohydrates (in grams) that are on the image you have selected. | Open-ended response |
| grapes 1 [if pasta1 = 1 or pasta4 $\neq$ .] | How often do you eat grapes? | 1. Rarely/Never 2. Occasionally 3. Often |
| grapes2 [if grapes1 = 2 or 3] | Select the image that matches the portion size you typically eat. If you typically eat a larger or smaller portion than any of the shown, select the image that comes closest. | 1. Portion size A 2. Portion size B 3. Portion size C 4. Portion size D 5. Portion size E 6. Portion size F |
| grapes3 [if grapes1 = 2 or 3] | A B C C F F | |
| grapes4 [if grapes2 ≠ .] | Type the amount of carbohydrates (in grams) that are on the image you have selected. | Open-ended response |
| bun1 [if grapes1 = 1 or grapes4 ≠ .] | How often do you eat wholegrain bread rolls? | 1. Rarely/Never 2. Occasionally 3. Often |
| bun2 [if bun1 = 2 or 3] | Select the image that matches the portion size you typically eat. If you typically eat a larger or smaller portion than any of the shown, select the image that comes closest. | 1. Portion size A 2. Portion size B 3. Portion size C 4. Portion size D 5. Portion size E |
| bun3 [if bun1 = 2 or 3] | A Vegt 40 g D E Vegt 100 g 140 g | |

| bun4 [if bun2 ≠ .] | Type the amount of carbohydrates (in grams) that are on the image | Open-ended |
|---|---|---|
| | you have selected. | response |

# 

| Scale/item [branching logic] | Question | Response categories |
|---|---|---|
| | about your satisfaction with your current insulin pum | p. Think about your |
| everyday life with the pump a | nd indicate the degree to which you agree or disagree | with the following |
| statements. | | |
| My insulin pump | | |
| idds1 | helps me to feel more in control of my diabetes | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds2 | works well when I need it | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds3 | does not really benefit me much | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds4 | helps me feel more positive about the future | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds5 | helps me to have good blood glucose control | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds6 | is too complicated | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds7 | is too much of a hassle to use | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds8 | has too many pieces and parts to manage | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds9 | takes too much time to use | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |

| | | 4. Agree |
|---|---|---|
| | | 5. Strongly agree |
| idds10 | is often embarrassing to use when I am in public | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds11 | makes it difficult to be as spontaneous as I'd like to | Strongly disagree |
| | be | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds12 | is inconvenient to use when I am away from home | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| idds13 | is a hassle to carry around | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |


| Scale/item [branching | Question | Response categories |
|---|---|---|
| logic] | | |
| _ | s concern your satisfaction with your current glucose meter | . – |
| blood glucose monitor or sensor). Base your answer on the meter you use the most or consider your primary | | |
| meter and indicate the degree to which you agree or disagree with the following statements. | | |
| devicetype | Please specify which glucose meter you are basing your | Sensor or Flash glucose |
| | answers on? | meter |
| | | 2. Blood sugar device |
| gmss_intro | My current blood glucose monitor/sensor | |
| gmss1 | helps me feel more satisfied with how things are going with my diabetes | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss2 | makes me think about diabetes more than I want to | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss3 | takes too much time to use | Strongly disagree |
| 8 | takes too mach time to use | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss4 | doesn't seem to be as accurate as I would like it to be | Strongly disagree 1. Strongly disagree |
| S11135-1 | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| amee5 | makes me worry a lot | Strongly disagree 1. Strongly disagree |
| gmss5 | makes me worry a for | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | 1 0 1 1 4 | 5. Strongly agree |
| gmss6 | is too much of a hassle to use | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss7 | gives me numbers that I don't entirely trust | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss8 | helps me feel less restricted by diabetes | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |

| | | 5. Strongly agree |
|---|---|---|
| gmss9 | makes me feel more frustrated with my diabetes | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss10 | helps me to be more spontaneous in daily life | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss11 | Causes too many skin irritations or bruises | Strongly disagree |
| | · | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss12 | often gives me results that don't make sense | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss13 | makes me feel more down and depressed | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss14 | helps me to be more open to new experiences in life | 1. Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |
| gmss15 | is too painful to use | Strongly disagree |
| | | 2. Disagree |
| | | 3. Neutral |
| | | 4. Agree |
| | | 5. Strongly agree |


| Scale/item [branching logic] | Question | Response categories |
|---|---|---|
| | how you experience wearing the insulin pump on your body. | .1 |
| bodyimageintro1 | Please indicate the degree to which you agree or disagree with the following statements: | |
| bodyimage1 | The insulin pump makes me feel me different in the eyes of others | <ol> <li>Strongly disagree</li> <li>Disagree</li> <li>Neither disagree</li> <li>nor agree</li> <li>Agree</li> <li>Strongly agree</li> </ol> |
| bodyimage2 | It bothers me that I always have an insulin catheter in my body | 1. Strongly disagree 2. Disagree 3. Neither disagree nor agree 4. Agree 5. Strongly agree |
| bodyimage3 | With the insulin pump, others immediately notice that I have diabetes | 1. Strongly disagree 2. Disagree 3. Neither disagree nor agree 4. Agree 5. Strongly agree |
| bodyimage4 | The insulin pump makes me less attractive | 1. Strongly disagree 2. Disagree 3. Neither disagree nor agree 4. Agree 5. Strongly agree |
| bodyimageintro2 | Please indicate the degree to which you agree or disagree with the following statements: | |
| bodyimage5 | The insulin pump bothers me when I sleep | <ol> <li>Strongly disagree</li> <li>Disagree</li> <li>Neither disagree</li> <li>agree</li> <li>Agree</li> <li>Strongly agree</li> </ol> |
| bodyimage6 | The insulin pump bothers me when I exercise | 1. Strongly disagree 2. Disagree 3. Neither disagree nor agree 4. Agree 5. Strongly agree |
| bodyimage7 | The insulin pump bothers me when I have sex | 1. Strongly disagree 2. Disagree 3. Neither disagree nor agree 4. Agree |

| | | 5. Strongly agree |
|---|---|---|
| bodyimage8 | The insulin pump prohibits me from wearing the clothes that I | 1. Strongly disagree |
| | want to wear | 2. Disagree |
| | | 3. Neither disagree |
| | | nor agree |
| | | 4. Agree |
| | | 5. Strongly agree |


| Scale/item<br>[branching | Question | Response categories |
|---|---|---|
| logic] | | |
| | we ask about your general health behavior, including exercise, diet and well as smoking status. | |
| exercise l | In a normal week, how much time do you spend doing physical activities that cause you to be short of breath (e.g., running, gymnastics, or ball games)? | 1. 0 minutes / No time 2. Less than 30 minutes 3. 30-60 minutes (0.5-1 hour) 4. 60-90 minutes (1- 1.5 hours) 5. 90-120 minutes (1.5-2 hours) 6. 120-150 minutes (2-2.5 hours) |
| | | 7. More than 150 minutes |
| exercise2 | In a normal week, how much time do you spend doing everyday exercise (e.g., walking, cycling or manual labor)? | 1. 0 minutes / No time 2. Less than 30 minutes 3. 30-60 minutes (0.5-1 hour) 4. 60-90 minutes (1- 1.5 hours) 5. 90-150 minutes (1.5-2.5 hours) 6. 150-300 minutes (2.5-5 hours) 7. More than 300 minutes (5 hours) |
| exercise3 | How much time do you spend sitting down on a regular day when sleep is not included? | 1. Pretty much all day 2. 13-15 hours 3. 10-12 hours 4. 7-9 hours 5. 4-6 hours 6. 1-3 hours 7. No time |
| diet1 | How many vegetables do you eat (raw or prepared)? Think in servings, e.g., a carrot or 100 g fried vegetables. If you eat both a carrot and 100 g of fried vegetables, you have eaten two servings. | 1. 6 a day or more 2. 5-6 a day 3. 3-4 a day 4. 1-2 a day 5. 5-6 a week 6. 3-4 a week 7. 1-2 a week |

| | | 8. Fewer or none |
|---|---|---|
| | | 6. Pewer of none |
| diet2 | How much fruit do you eat? | 1. 6 a day or more |
| | | 2. 5-6 a day |
| | Think in servings, e.g., an apple or 10 grapes. | 3. 3-4 a day |
| | | 4. 1-2 a day |
| | | 5. 5-6 a week |
| | | 6. 3-4 a week |
| | | 7. 1-2 a week |
| | | 8. Fewer or none |
| diet3 | How often do you eat whole grains? | 1. More than 2 |
| | | times a day |
| | Whole grain foods include, e.g., oatmeal, rye bread, whole grain bread or | 2. 1-2 times a day |
| | whole grain pasta. | 3. 4-6 times a week |
| | | 4. 1-3 times a week |
| | | 5. Rarely or never |
| diet4 | How often do you eat fish (fresh, prepared, or canned)? | 1. More than once a |
| | | day |
| | | 2. 5-7 times a week |
| | | 3. 3-4 times a week |
| | | 4. 1-2 times a week |
| | | 5. Rarely or never |
| diet5 | Do you follow The Danish Health Authority's recommendation to eat less | 1. Almost always |
| | saturated fat and choose plant oil instead? | 2. Usually |
| | | 3. Occasionally |
| | Recommendation: Choose lean meat and lean dairy products, and limit | 4. Rarely |
| | the amount of butter, | 5. Never |
| | whole-fat cheeses and cream. Use plant oil/liquid margarine in cooking. | |
| diet6 | To the best of your knowledge, how often does is your intake of fast | 1. Never or very |
| | carbohydrates in the form of, e.g., candy, cake, ice cream and other | rarely |
| | sweets so great that it causes a prolonged blood sugar increase? | 2. Rarely (about |
| | | once a month) |
| | | 3. Occasionally (a |
| | | few times a month) |
| | | 4. Often (1-2 times |
| | | a week) |
| | | 5. Very often (daily |
| | | or almost daily) |
| alcohol | How much beer, wine, and/or spirits do you drink on average per week? | 1. I do not drink |
| | Please reply in units of alcohol (1 unit equals, e.g., 1 beer, 1 glass of | 2. 1-7 units |
| | wine, 1 schnapps or 1 shot). | 3. 8-14 units |
| | | 4. 14-21 units |
| | | 5. More than 21 |
| | | units |
| smoking | Do you smoke? | 1. No |
| | | 2. Yes, daily |
| | | 3. Yes, occasionally |
| | | 4. Former smoker |


| Scale/item | Question | Response |
|---|---|---|
| [branching logic] | | categories |
| - | e about low blood sugars. We would like to stress that your responses to the | e following |
| hypobehavior_intro | Here are five statements about things people with diabetes sometimes do to | |
| | avoid low blood sugar and consequences of it. Please specify what you | |
| | have done the last month in your everyday life to AVOID low blood sugar and its effects. | |
| | To avoid low blood sugar and the repercussions of it, I have | |
| hypob1 | limited my out of town travel | 1. Never |
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| | | always |
| hypob2 | avoided visiting friends | 1. Never |
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| | | always |
| hypob3 | made sure there were other people around | 1. Never |
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| | | always |
| hypob4 | kept my blood sugar higher than usual in social situations | 1. Never |
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| | | always |
| hypob5 | kept my blood sugar higher than usual while doing important tasks | 1. Never |
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| 1 | How we design the design of th | always |
| hypoworry_intro | Here are six statements about concerns that people with diabetes sometimes have due to low blood sugar. | |
| | Please indicate how often during the past month you have been | |
| | CONCERNED about each statement due to low blood sugar. | |
| | Because my blood sugar could drop, I was worried about | |

| hypow1 | not to recognizing I was having a low blood sugar | 1. Never |
|---|---|---|
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| | | always |
| hypow2 | passing out in public | 1. Never |
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| | | always |
| hypow3 | having a hypoglycemic episode while driving | 1. Never |
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| | | always |
| hypow4 | low blood glucose interfering with important things I was doing | 1. Never |
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| | | always |
| hypow5 | becoming hypoglycemic during sleep | 1. Never |
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| | | always |
| hypow6 | getting emotionally upset and difficult to deal with | 1. Never |
| | | 2. Rarely |
| | | 3. Sometimes |
| | | 4. Often |
| | | 5. Almost |
| | | always |


| Scale/item | Question | Response categories |
|---|---|---|
| [branching logic] | | |
| Below is a list of statements about various forms of concern that many people with type 1 diabetes experience. | | |
| We ask you to assess the past month. | the extent to which each of the following statements has been a pr | roblem for you within |
| dds1 | Feeling that I am not as skilled at managing diabetes as I should be | <ol> <li>Not a problem</li> <li>A slight problem</li> <li>A moderate problem</li> <li>A somewhat serious problem</li> <li>A serious problem</li> <li>A very serious problem</li> </ol> |
| dds2 | Feeling that I don't eat as carefully as I probably should | <ol> <li>Not a problem</li> <li>A slight problem</li> <li>A moderate problem</li> <li>A somewhat serious problem</li> <li>A serious problem</li> <li>A very serious problem</li> </ol> |
| dds3 | Feeling that I don't notice the warning signs of hypoglycemia as well as I used to | <ol> <li>Not a problem</li> <li>A slight problem</li> <li>A moderate problem</li> <li>A somewhat serious problem</li> <li>A serious problem</li> <li>A very serious problem</li> </ol> |
| dds4 | Feeling that people treat me differently when they find out I have diabetes | <ol> <li>Not a problem</li> <li>A slight problem</li> <li>A moderate problem</li> <li>A somewhat serious problem</li> <li>A serious problem</li> <li>A very serious problem</li> </ol> |
| dds5 | Feeling discouraged when I see high blood glucose numbers that I can't explain | <ol> <li>Not a problem</li> <li>A slight problem</li> <li>A moderate problem</li> <li>A somewhat serious problem</li> <li>A serious problem</li> <li>A very serious problem</li> </ol> |
| dds6 | Feeling that my family and friends make a bigger deal out of diabetes than they should | Not a problem A slight problem |

| | | 2. A mandamet a martal. |
|---|---|---|
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds7 | Feeling that I can't tell my diabetes doctor what is really on my | 1. Not a problem |
| | mind | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds8 | Feeling that I am not taking as much insulin as I should | 1. Not a problem |
| | | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds9 | Feeling that there is too much diabetes equipment and stuff I | 1. Not a problem |
| | must always have with me | 2. A slight problem |
| | must arways have with me | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds10 | Feeling like I have to hide my diabetes from other people | 1. Not a problem |
| dusto | recting like I have to finde my diabetes from other people | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds11 | Eagling that my friends and family warms many shout | 1. Not a problem |
| uusii | Feeling that my friends and family worry more about | _ |
| | hypoglycemia than I want them to | 2. A slight problem |
| | | 3. A moderate problem 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| 44.45 | | problem |
| dds12 | Feeling that I don't check my blood glucose level as often as I | 1. Not a problem |
| | probably should | 2. A slight problem |
| | | 3. A moderate problem |

| | | 4. A somewhat serious |
|---|---|---|
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds13 | Feeling worried that I will develop serious long-term | 1. Not a problem |
| ddS13 | complications, no matter how hard I try | 2. A slight problem |
| | complications, no matter now hard I dy | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds14 | Facility 4ha4 I dow/44 halls I walle was different way dishada | • |
| ddS14 | Feeling that I don't get help I really need from my diabetes | 1. Not a problem |
| | doctor about managing diabetes | 2. A slight problem |
| | | 3. A moderate problem 4. A somewhat serious |
| | | problem |
| | | <ul><li>5. A serious problem</li><li>6. A very serious</li></ul> |
| | | problem |
| dds15 | Fasting frightened that I could have a goviere home abreautic | * |
| aasis | Feeling frightened that I could have a serious hypoglycemic | 1. Not a problem |
| | event when I'm asleep | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| 11.16 | | problem |
| dds16 | Feeling that thoughts about food and eating control my life | 1. Not a problem |
| | | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| 11.15 | | problem |
| dds17 | Feeling that my friends or family treat me as if I were more | 1. Not a problem |
| | fragile or sicker than I really am | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| 11.10 | | problem |
| dds18 | Feeling that my diabetes doctor doesn't really understand what | 1. Not a problem |
| | it's like to have diabetes | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |

| | | 16.4 |
|---|---|---|
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds19 | Feeling concerned that diabetes may make me less attractive to | 1. Not a problem |
| | employers | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds20 | Feeling that my friends or family act like "diabetes police" | 1. Not a problem |
| | (bother me too much) | 2. A slight problem |
| | (************************************** | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds21 | Faciling that I've get to be perfect with my dishetes management | 1. Not a problem |
| dusz i | Feeling that I've got to be perfect with my diabetes management | • |
| | | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds22 | Feeling frightened that I could have a serious hypoglycemic | 1. Not a problem |
| | event while driving | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds23 | Feeling that my eating is out of control | 1. Not a problem |
| | | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds24 | Feeling that people will think less of me if they knew I had | 1. Not a problem |
| | diabetes | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 5.11 Serious problem |

| | | 6. A very serious |
|---|---|---|
| | | problem |
| dds25 | Feeling that no matter how hard I try with my diabetes, it will | 1. Not a problem |
| | never be good enough | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds26 | Feeling that my diabetes doctor doesn't know enough about | 1. Not a problem |
| | diabetes and diabetes care | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds27 | Feeling that I can't ever be safe from the possibility of a serious | 1. Not a problem |
| | hypoglycemic event | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds28 | Feeling that I don't give my diabetes as much attention as I | 1. Not a problem |
| | probably should | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |
| dds29 | Feeling that I can't do my job because of my diabetes | 1. Not a problem |
| | | 2. A slight problem |
| | | 3. A moderate problem |
| | | 4. A somewhat serious |
| | | problem |
| | | 5. A serious problem |
| | | 6. A very serious |
| | | problem |


| Scale/item | Question | Response categories |
|---|---|---|
| [branching logic] | | |
| How supportive hav | How supportive have the following people been in helping you to manage your diabetes in the past month? | |
| sos1 | Your family | 1. Not supportive |
| | | 2. Somewhat supportive |
| | | 3. Very supportive |
| | | 4. Do not have these (not relevant |
| | | with support from here) |
| sos2 | Friends or other people close to you | 1. Not supportive |
| | | 2. Somewhat supportive |
| | | 3. Very supportive |
| | | 4. Do not have these (not relevant |
| | | with support from here) |
| sos3 | People at your place of work or study | 1. Not supportive |
| | | 2. Somewhat supportive |
| | | 3. Very supportive |
| | | 4. Do not have these (not relevant |
| | | with support from here) |
| sos4 | Your diabetes healthcare provider | 1. Not supportive |
| | | 2. Somewhat supportive |
| | | 3. Very supportive |
| | | 4. Do not have these (not relevant |
| | | with support from here) |
| sos5 | Other people with type 1 diabetes | 1. Not supportive |
| | | 2. Somewhat supportive |
| | | 3. Very supportive |
| | | 4. Do not have these (not relevant |
| | | with support from here) |
| sos6 | People on social media (e.g. in Facebook groups | 1. Not supportive |
| | for people with type 1 diabetes) | 2. Somewhat supportive |
| | | 3. Very supportive |
| | | 4. Do not have these (not relevant |
| | | with support from here) |


| Scale/item [branching | Question | Response |
|---|---|---|
| logic] | | categories |
| • | ou perceive your own abilities to do and achieve the things you war | nt to |
| in your life with diabetes | s. | |
| | ree the following statements fit you. | |
| selfeffi1 | I can always manage to solve difficult problems if I try hard | 1. Not at all true |
| | enough | 2. Hardly true |
| | | 3. Moderately true |
| | | 4. Exactly true |
| selfeffi2 | If someone opposes me, I can find the means and ways to get what | 1. Not at all true |
| | I want | 2. Hardly true |
| | | 3. Moderately true |
| | | 4. Exactly true |
| selfeffi3 | It is easy for me to stick to my aims and accomplish my goals | 1. Not at all true |
| | | 2. Hardly true |
| | | 3. Moderately true |
| | | 4. Exactly true |
| selfeffi4 | I am confident that I could deal efficiently with unexpected events | 1. Not at all true |
| | | 2. Hardly true |
| | | 3. Moderately true |
| | | 4. Exactly true |
| selfeffi5 | Thanks to my resourcefulness, I know how to handle unforeseen | 1. Not at all true |
| | situations | 2. Hardly true |
| | | 3. Moderately true |
| | | 4. Exactly true |
| selfeffi6 | I can solve most problems if I invest the necessary effort | 1. Not at all true |
| | | 2. Hardly true |
| | | 3. Moderately true |
| | | 4. Exactly true |
| selfeffi7 | I can remain calm when facing difficulties because I can rely on | 1. Not at all true |
| | my coping abilities | 2. Hardly true |
| | , | 3. Moderately true |
| | | 4. Exactly true |
| selfeffi8 | When I am confronted with a problem, I can usually find several | 1. Not at all true |
| Selicino | solutions | 2. Hardly true |
| | SOLUTIONS | 3. Moderately true |
| | | 4. Exactly true |
| selfeffi9 | If I am in trouble, I can usually think of a solution | 1. Not at all true |
| SCHOHI) | 11 1 dill ill trouble, I call usually tillik of a solution | 2. Hardly true |
| | | 3. Moderately true |
| | | 4. Exactly true |
| selfeffi10 | I can usually handle whatever comes my way | 1. Not at all true |
| SCHEIHIU | i can usuany nandie whatever comes my way | |
| | | 2. Hardly true |
| | | 3. Moderately true |
| | | 4. Exactly true |

# 

| Scale/item | Question | Response categories |
|---|---|---|
| [branching logic] | | |
| Long-term blood glu | Long-term blood glucose (HbA1c) | |
| hba1c_intro | What long-term blood sugar level (HbA1c) would | 1. % |
| | you yourself like to be at? You can enter your | 2. mmol/mol |
| | answer in either % or mmol/mol by indicating your | 3. I have not set myself a fixed |
| | preference here. | goal for HbA1c |
| hba1c_goal_percent | HbA1c (%) | Open-ended response |
| [if hba1c_intro = 1] | | |
| hba1c_goal_mmol | HbA1c (mmol/mol) | Open-ended response |
| [if hba1c_intro = 2] | | |
| hba1c_realistic [if | How likely do you think it is that you will have | 0. Completely unlikely |
| hba1c_intro $\neq 3$ ] | achieved/stayed on that particular long-term blood | 10. Completely likely |
| | sugar level (HbA1c) in a year? Please indicate your | |
| | answer on a scale from 0-10. | |


| Scale/item [branching logic] | Question | Response categories |
|---|---|---|
| | are more about your general health and overall satisfaction with life. | |
| healthstatus | How good or bad do you consider your health today? Please indicate your answer on a scale from 0-10. | 0. Very bad<br>10. Very good |
| satisfaction | How satisfied are you with your life today all things considered? Please indicate your answer on a scale from 0-10. | 0. Not at all satisfied 10. Completely satisfied |
| who5_intro | Please indicate for each of the 5 statements which is closest to how you have been feeling over the past 2 weeks. | |
| | Over the past 2 weeks | |
| who51 | I have felt cheerful and in good spirits | 1. All of the time 2. Most of the time 3. More than half the time 4. Less than half the time 5. Some of the time 6. At no time |
| who52 | I have felt calm and relaxed | 1. All of the time 2. Most of the time 3. More than half the time 4. Less than half the time 5. Some of the time 6. At no time |
| who53 | I have felt active and vigorous | 1. All of the time 2. Most of the time 3. More than half the time 4. Less than half the time 5. Some of the time 6. At no time |
| who54 | I woke up feeling fresh and rested | 1. All of the time 2. Most of the time 3. More than half the time 4. Less than half the time 5. Some of the time 6. At no time |
| who55 | my daily life has been filled with things that interest me | 1. All of the time |

| 2. Most of the time |
|---------------------|
| 3. More than half |
| the time |
| 4. Less than half |
| the time |
| 5. Some of the time |
| 6. At no time |

# 

| Scale/item | Question | Response |
|---|---|---|
| [branching logic] | | categories |
| | ndemic may impact the lives and opportunities of insulin pump users in r | elation to |
| treatment and educ | cation. | |
| covid19_intro | How is the COVID-19 pandemic CURRENTLY impacting the following aspects of your life? | |
| covid1 | Your diabetes Your diabetes | 1. Very negative impact 2. Negative impact 3. Slightly negative impact 4. No impact 5. Slightly positive impact 6. Very positive impact |
| covid2 | Your sleep | 7. Not applicable 1. Very negative |
| covid3 | Your physical health | impact 2. Negative impact 3. Slightly negative impact 4. No impact 5. Slightly positive impact 6. Very positive impact 7. Not applicable 1. Very negative |
| COVID | Tour physical nearth | impact 2. Negative impact 3. Slightly negative impact 4. No impact 5. Slightly positive impact 6. Very positive impact 7. Not applicable |
| covid4 | Your emotional wellbeing | 1. Very negative impact 2. Negative impact |

| | | 2 01:-1-4 |
|---|---|---|
| | | 3. Slightly |
| | | negative impact |
| | | 4. No impact |
| | | 5. Slightly |
| | | positive impact |
| | | 6. Very positive |
| | | impact |
| | | 7. Not applicable |
| covid5 | Your financial situation | 1. Very negative |
| | | impact |
| | | 2. Negative |
| | | impact |
| | | 3. Slightly |
| | | negative impact |
| | | 4. No impact |
| | | 5. Slightly |
| | | positive impact |
| | | 6. Very positive |
| | | impact |
| | | 7. Not applicable |
| covid6 | Your relationship with your family, friends and peers | 1. Very negative |
| | 1 3 | impact |
| | | 2. Negative |
| | | impact |
| | | 3. Slightly |
| | | negative impact |
| | | 4. No impact |
| | | 5. Slightly |
| | | positive impact |
| | | 6. Very positive |
| | | impact |
| | | 7. Not applicable |
| covid7 | Your leisure activities | 1. Very negative |
| Covidy | 1 our resource detrivities | impact |
| | | 2. Negative |
| | | impact |
| | | 3. Slightly |
| | | negative impact |
| | | 4. No impact |
| | | 5. Slightly |
| | | positive impact |
| | | 6. Very positive |
| | | impact |
| | | 7. Not applicable |
| covid8 | Your work or studies | 1. Very negative |
| COVIGO | 1 our work or studies | |
| | | impact |
| | | 2. Negative |
| | | impact |
| | | 3. Slightly |
| | | negative impact |

| | | 4. No impact |
|---|---|---|
| | | 5. Slightly |
| | | positive impact |
| | | 6. Very positive |
| | | impact |
| | | 7. Not applicable |
| covid9 | Your feelings about the future | 1. Very negative |
| | | impact |
| | | 2. Negative |
| | | impact |
| | | 3. Slightly |
| | | negative impact |
| | | 4. No impact |
| | | 5. Slightly |
| | | positive impact |
| | | 6. Very positive |
| | | impact |
| | | 7. Not applicable |
| covidrisk | How likely do you think it is for you to be become seriously ill if you get | 0. Completely |
| | infected with the COVID-19 virus? Please indicate your answer on a | unlikely |
| | scale from 0-10. | 10. Completely |
| | | likely |

# 

| Scale/item | Question | Response |
|---|---|---|
| [branching | | categories |
| logic] | | |
| You are now f | nished with the part of the questionnaire about your diabetes and your insu | ilin pump. |
| to these question | lso want to answer the next questions, which are more about you in general ons will be used to gain an understanding of how people make decisions. are not a test and there are no right or wrong answers. | terms. Four unswer |
| lottery | Imagine that you unexpectedly inherit 2,500 kr from a distant relative. You | 1. I choose to |


| Scale/item | Question | Response |
|---|---|---|
| [branching logic] | | categories |
| Where do you stand | with regards to taking risks? | |
| risk1 | Are you someone who is willing to take risks in general? Please indicate | 0. Fully |
| | your answer on a scale from 0-10. | unwilling |
| | | 10. Fully |
| | | willing |
| risk2 | Are you someone who is willing to take risks with your health in | 0. Fully |
| | general? Please indicate your answer on a scale from 0-10. | unwilling |
| | | 10. Fully |
| | | willing |
| risk3 | Are you someone who is willing to take risks with your financial | 0. Fully |
| | situation? Please indicate your answer on a scale from 0-10. | unwilling |
| | | 10. Fully |
| | | willing |

# 

| Scale/item | Question | Response |
|---|---|---|
| [branching logic] | | categories |
| How patient and im | ipulsive are you? | |
| patience | In general, how patient are you? Please indicate your answer on a scale | 0. Very |
| | from 0-10. | impatient |
| | | 10. Very patient |
| impulsive | Are you a person who generally acts impulsively, or do you think a lot | 0. Not impulsive |
| | about things before you act? Please indicate your answer on a scale from | at all |
| | 0-10. | 10. Very |
| | | impulsive |
| riskage | Think about the future. How likely do you think it is that you will | 0. Completely |
| | experience your 90th birthday? Please indicate your answer on a scale from | unlikely |
| | 0-10. | 10. Completely |
| | | likely |


| Scale/item [branching logic] | Question | Response categories |
|---|---|---|
| liveplando_intro | To what degree do you agree with the following statements? | |
| livelife | I live life one day at a time and do not think too much about my future | <ol> <li>Strongly disagree</li> <li>Disagree</li> <li>Neither disagree nor agree</li> <li>Agree</li> <li>Strongly agree</li> </ol> |
| planlife | I plan everything in good time | <ol> <li>Strongly disagree</li> <li>Disagree</li> <li>Neither disagree nor agree</li> <li>Agree</li> <li>Strongly agree</li> </ol> |
| dolife | When I set a goal for myself, I always achieve it | <ol> <li>Strongly disagree</li> <li>Disagree</li> <li>Neither disagree nor agree</li> <li>Agree</li> <li>Strongly agree</li> </ol> |


| Scale/item | Question | Response |
|---|---|---|
| [branching logic] | | categories |
| The following qu | estions are about time and money. | |
| TD1 4* | | |
| The questions are | e not a test and there are no right or wrong answers. | |
| priselist_intro1 | Imagine that you can choose between getting 5,000 kr. today or another | |
| prisenst_intro1 | amount in 1 year. What amount do you prefer in each of the following seven | |
| | situations? The money is yours no matter what, and there is no risk of you | |
| | losing a future amount if you choose to wait. | |
| | losing a ratare amount if you encose to wait. | |
| | We have filled out the first answer for you as we believe you would prefer to | |
| | have 5,000 kr. in your hand today rather than in 1 year. | |
| pricelist1 | , | 1. 5,000 kr. |
| • | | today |
| | | 2. 5,000 kr. |
| | | in a year |
| pricelist2 | | 1. 5,000 kr. |
| | | today |
| | | 2. 5,100 kr. |
| | | in a year |
| pricelist3 | | 1. 5,000 kr. |
| | | today |
| | | 2. 5,250 kr. |
| | | in a year |
| pricelist4 | | 1. 5,000 kr. |
| | | today |
| | | 2. 5,500 kr. |
| | | in a year |
| pricelist5 | | 1. 5,000 kr. |
| | | today |
| | | 2. 6,000 kr. |
| | | in a year |
| pricelist6 | | 1. 5,000 kr. |
| | | today |
| | | 2. 7000 kr. in |
| | | a year |
| pricelist7 | | 1. 5,000 kr. |
| | | today |
| | | 2. 9000 kr. in |
| | | a year |

## 

| Scale/item | Question | Response |
|-------------------|----------|------------|
| [branching logic] | | categories |

The next questions are like the previous, only now the time horizon varies.

How much would you require in addition to the 5,000 kr. to wait for the money in each scenario?

There are no right or wrong answers.

When you enter an amount, the total sum is calculated in the following field, and you therefore do not have to write anything in this field.

| write anything in this | , neru. | |
|---|---|---|
| tp1 | How much money would you require in addition to the 5,000 kr. if you | Open-ended |
| | had to wait 1 month to get the money? | response |
| $tp1\_calc [if tp1 \neq .]$ | This means that instead of 5,000 kr. today, you will get | X kr. in 1 month |
| tp2 | Against waiting 3 months? | Open-ended |
| | | response |
| $tp2$ _calc [if $tp2 \neq .$ ] | This means that instead of 5,000 kr. today, you will get | X kr. in 3 |
| | | months |
| tp3 | Against waiting 6 months? | Open-ended |
| | | response |
| tp3_calc [if tp3 $\neq$ .] | This means that instead of 5,000 kr. today, you will get | X kr. in 6 |
| | | months |
| tp4 | Against waiting 12 months? | Open-ended |
| | | response |
| $tp4$ _calc [if $tp4 \neq .$ ] | This means that instead of 5,000 kr. today, you will get | X kr. in 12 |
| | | months |
| tp5 | Against waiting 24 months? | Open-ended |
| | | response |
| $tp5$ _calc [if $tp5 \neq .$ ] | This means that instead of 5,000 kr. today, you will get | X kr. in 24 |
| | | months |

# 

| Scale/item [branching logic] | Question | Response categories |
|---|---|---|
| Now imagine a situation where you cannot get the 5,000 kr. before 12 months from now. | | |
| tp24 | How much money would you require in addition to the 5,000 kr. in 12 months for you to wait another 12 months to get the money? | Open-ended response |
| tp24_calc | This means that instead of getting 5,000 kr. in 12 months you will get | X kr. in 24<br>months |


| Scale/item [branching | Question | Response categories |
|---|---|---|
| logic] | | |
| Thank you so much for | your help! | |
| | to learn more about how people with type 1 diabetes use a<br>knowledge to improve treatment options for insulin pump | |
| Hospital Hillerød and S | teno Diabetes Center Copenhagen. | |
| sdeenoh | Are you treated at Nordsjællands Hospital Hillerød or<br>Steno Diabetes Center Copenhagen? | Nordsjællands Hospital Hillerød Steno Diabetes Center Copenhagen |
| contact | Can we send you a similar questionnaire in a year? | 1. Yes<br>2. No |
| panel | At Steno Diabetes Center Copenhagen, we carry out numerous research projects with different research subjects on an ongoing basis. In the context of this, we have been given permission to create a register of people interested in participating in new research projects. By ticking here, you agree that we may contact you with information about the possibility of participation in upcoming research projects/trials. Your consent is valid for 1 year. You can say no to participating in the trials at any time, just as you can always withdraw your consent to be included in the register. | 1. Yes, I would like to be included in the register and contacted via e-Boks when new research projects come in 2. Yes, I would like to be included in the register and contacted via e-Boks and/or phone when new research projects come in. 3. I do not want to be part of the register |
| phone [if panel = 2] | Please provide a phone number we may contact you at. Enter only the 8 digits. | Open-ended response. |
| carbcountanswer_intro | Bonus info: fact list for the carbohydrate counting exercise! | |
| carbcountanswer1 | Chocolate: You replied that there are [choco4] grams of carbohydrates in the chocolate in the selected image. The exact amount of carbohydrates is: | X |
| carbcountanswer2 | Pasta: You replied that there is [pasta4] grams of carbohydrates in the pasta in the selected image. The exact amount of carbohydrates is: | X |
| carbcountanswer3 | Grapes: You replied that there are [grapes4] grams of carbohydrates in the grapes in the selected image. The exact amount of carbohydrates is: | X |
| carbcountanswer4 | Buns: You replied that there are [bun4] grams of carbohydrates in the bread roll on the selected image. The exact amount of carbohydrates is: | X |